CLINICAL TRIAL: NCT06998316
Title: Linguistical Validation of a Spondylo-arthritis Screening Tool for Patients Suffering From Inflammatory Bowel Disease
Brief Title: Spondylo-arthritis Screening Tool Among Patient Suffering From Inflammatory Bowel Disease
Acronym: QUESAM
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinique des Cèdres, Echirolles (Unknown)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0348
Record Dates: First submitted 2025-05-12; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Spondylarthritis; Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Spondylitis, Ankylosing
Keywords: spondylarthritis; Crohn Disease; Ulcerative Colitis; Inflammatory Bowel Diseases; screening tools
MeSH Terms: conditions — Spondylarthritis; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People with inflammatory bowel disease: Patient followed in gastro-enterology for an inflammatory bowel disease. These represent every-patient in our study.
  Interventions: Other: Screening questionnaire

INTERVENTIONS:
Other: Screening questionnaire — Every patient will answer the 2 screening questionnaires given to them, once at baseline and a second time after 1 month.

SUMMARY:
The QUESAM study aims to translate into French and validate the traduction of 2 screening questionnaires for spondylo-arthritis among people with inflammatory bowel disease.

DETAIL (DETection of Arthritis in Inflammatory boweL diseases) and IBIS-Q (Inflammatory Bowel disease Identification of Spondyloarthritis Questionnaire) questionnaires are built to determine which patients might benefit from a rheumatologic consultation, for a potential rheumatologic inflammatory disease.

The investigators will translate the 2 questionnaire in french thanks to an external translation company, from english to french, then back to english to make sure the translation is correct.

Then, the main question is:

is there a conceptual and semantic equivalence beetween the original english questionnaire and the french-translated one.

Participant will answer the 2 screening questionnaire, one initial time during a consultation, and a second time after 1 month.

DETAILED DESCRIPTION:
This is not an actual interventionnal or observationnal study. Investigators will try to provide a statistical validation of 2 questionnaires on people followed in gastro-enterology for an inflammatory bowel disease.

In the first place, investigators will translate the 2 questionnaires

* "The DETection of Arthritis in Inflammatory boweL diseases (DETAIL) questionnaire: development and preliminary testing of a new tool to screen patients with inflammatory bowel disease for the presence of spondyloarthritis, Di Carlo et al (2017)"
* "The IBIS-Q [IBd Identification of Spondyloarthritis Questionnaire]: A Novel Tool to Detect Both Axial and Peripheral Arthritis in Inflammatory Bowel Disease Patients, Variola et al (2020) From english to french, with a specialized company in scientific translation.

Investigators will then, with the help of 5 patients, determine if the translated final version is easy to understand, and eventually adjust the questionnaires if needed.

If a modification is needed, 5 other patients will be reached to look for any unclear formulation.

If no modification is needed, the questionnaire will be given to eligible patients until 200 answers are reached. People will be recruited during a standard care consultation or a one day-hospitalization for biological treatment

Invistigators will, on top of the questionnaires, be collecting the

* sex
* age
* study level
* type of inflammatory bowel disease
* presence of musculoskeletal pain
* duration of articulary and bowel disease
* previous treatment by biologic
* known spondylo-arthritis

At 1 month, participants will be contacted by mail, so that they fill the questionnaires again.

At last, with the answers to the 400 hundreds questionnaires (200 patients, baseline questionnaire + the one month reminder), investigators will be able to make the statistic analyzes required for the statistical validation of the questionnaires, in french.

Outside of the statistical validation, if the questionnaire are in favor of a rheumatologic disease, the gastro-enterologist can address patients to a rheumatology department.

General praticionner will then receive a report of the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an inflammatory bowel disease according to gastroenterologist

Exclusion Criteria:

* No exclusion criteria
* Difficulty for understanding or reading french
* Persons covered by articles L1121-5 to L1121-8 of the French Public Health Code
* Patients with no social security coverage.
* Patients refusing to participate voluntarily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is people with inflammatory bowel disease
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
translation and cross-cultural adaptation in french of the questionnaires developped by Di Marco et al (2017) and Variola et al (2020) | 13 months
  This is a composite criterion combining conceptual equivalence and semantic equivalence of items between the transcultural adaptation of the scale and its original version. Conceptual equivalence will be judged on the results of factorial analysis (exploratory and confirmatory). Semantic equivalence of items will be based on evaluation by a panel of experts.

SECONDARY OUTCOMES:
acceptability of the instrument via the proportion of missing data for each item | Baseline and one month later
Evaluation of the internal consistency assessed by the average inter-item correlation, the average item-result correlation and cronbach's alpha coefficient | baseline and one month later
  These tests aim to determine if the different items are close enough to measure the same thing and still different enough not to be redundant.
evaluation of the reliability of the questionnaire through an intra-rater reliability with the intra-class correlation. | Baseline and one month later
  Aims to determine if one rater answers the same questions the same way at two different moments.
Comparaison of the acceptability of the instrument via the proportion of missing data for each item | 13 months
  this will be done by comparing the proportion of missing data for the 2 questionnaires
Comparaison of internal consistency of the 2 questionnaires | 13 months
  Through the comparaison of the average inter-item correlation, the average item-result correlation and cronbach's alpha coefficient
Comparaison of reliability of the 2 questionnaire | 13 months
  Through comparaison of an intra-rater reliability with the intra-class correlation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No